CLINICAL TRIAL: NCT03939364
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled, Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of SBS-101 After Intraoral Application in Patients With Oral Premalignant Lesions (OPL)
Brief Title: This Study is to Evaluate the Safety and Pharmacokinetics of SBS-101 in Patients With Oral Premalignant Lesions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Delays due to manufacturing and the COVID-19 pandemic
Sponsor: Skyline Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SBS-101-CL-001
Record Dates: First submitted 2019-04-18; First posted 2019-05-06 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Leukoplakia, Oral
Keywords: Erythroplakia, oral; Erythro-leukoplakia, oral
MeSH Terms: conditions — Leukoplakia, Oral; Erythroplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.1% SBS-101 (Experimental)
  Interventions: Drug: SBS-101
- 0.3% SBS-101 (Experimental)
  Interventions: Drug: SBS-101
- 0.2% SBS-101 (Experimental)
  Interventions: Drug: SBS-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SBS-101 — Isotretinoin Oral-Adhesive Film
  Arms: 0.1% SBS-101; 0.2% SBS-101; 0.3% SBS-101
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will be the first study investigating the safety, pharmacokinetics (PK), and efficacy of SBS-101 on oral pre-malignant lesions. As such, no clinical data has yet been generated using SBS-101 oral adhesive film.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to comprehend and willing to sign an Informed Consent Form.
2. Patient is willing and able to follow all study instructions and to attend all study visits
3. Patient is male or female aged 18 years or older at Screening.
4. Patient has oral leukoplakia or erythroplakia at least 5mm in length on its longest axis with histopathology showing mild, moderate, or severe dysplasia (index lesion histology score of ≥2) with incisional (punch) biopsy at Screening (or within 30 days prior to Screening).
5. Patient agrees to not use any topical therapies (i.e. use of over the counter and medically prescribed topical creams, ointments, or oral rinses) on the index lesion other than the study drug that, in the Investigator's opinion, might influence the status of the index lesion for the duration of the study.
6. Patient agrees to not apply any other topical products or use potential irritants (i.e. alcohol containing mouthwash) to the oral premalignant lesions throughout the study. Note: mouthwash that includes non-alcohol containing formulations of Listerine and Crest is acceptable to use during the study.
7. If female, patient is non-pregnant, non-lactating and is not planning for pregnancy during the study period or for 1 month after the last dose of study drug.
8. Female patients of non-childbearing potential must meet the following requirements:

   1. Pre-menopausal with documentation of surgical sterilization (i.e., hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or bilateral salpingectomy) at least 3 months prior to study entry.
   2. Post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with follicle-stimulating hormone (FSH) level ≥40 milli-international units per milliliter (mIU/mL) at Screening.
9. Female patients of child-bearing potential must select and commit to use 2 forms of effective contraception simultaneously, at least 1 of which must be a primary form, unless absolute abstinence is the chosen method, or the patient has undergone a hysterectomy. Patients must use 2 forms of effective contraception at least 1 month prior to study initiation (Screening), during the study, and for 1 month after the final dose of study drug.

   Primary (hormonal or surgical)
   1. Tubal ligation
   2. Partner's vasectomy
   3. Intrauterine devices
   4. Birth control pills
   5. Injectable/implantable/insertable hormonal birth control products Secondary (Barrier Method)

   <!-- -->

   1. Diaphragm (with spermicide)
   2. Cervical cap (with spermicide)
   3. Male condom (with spermicide)
10. Male patients must agree to use condoms during sexual intercourse during the study and for 3 months after the final dose of study drug. If a female partner is of childbearing potential, she should use contraception as detailed in Inclusion criterion

    # 9. Males must also agree to not donate sperm from the time of first dosing and for 3 months after the final dose of study drug.
11. Patient's Eastern Cooperative Oncology Group (ECOG) performance status grade is 0 or 1 at Screening.
12. Patient's organ function is determined to be adequate based on laboratory testing at Screening (e.g. Hemoglobin levels ≥ 10g/dl; White Blood Cells (WBC) ≥ 3,000/μL; Platelets ≥ 100,000/μL; Total bilirubin ≤ 1.5x Upper Limit of Normal (ULN); Aspartate Aminotransferase (AST)/ Alanine aminotransferase (ALT) < 2x Upper Limit of Normal (ULN);, Blood urea nitrogen (BUN) & serum creatinine ≤ 1.5x Upper Limit of Normal (ULN); Lactate dehydrogenase (LDH) ≤ 1.5x Upper Limit of Normal (ULN); Glucose < 200 mg/dL; Thyroid Stimulating Hormone (TSH) ≤ 5.0 μU/mL; C-Reactive Protein < 5.0 mg/L).
13. Negative urine drug screen at Screening.
14. Patient is in good general health and free of any known disease state or physical condition which, in the Investigator's opinion, might impair evaluation of the oral premalignant lesions or which exposes the patient to an unacceptable risk by participating in the study.

Exclusion Criteria:

1. Patient has oral lesions to be treated that are infected (e.g. lesions that require local or systemic antimicrobial, antifungal, or antiviral therapy to treat an infection) within 14 days of Randomization.
2. Patients must not use any systemic (e.g., oral or injectable) corticosteroid therapy during the study or within 30 days prior to Screening. However, use of topical, inhaled, ophthalmic, intraarticular and intralesional steroids is permitted.
3. Patient has used any topical or systemic chemotherapeutic product within 30 days prior to Randomization.
4. Use of smokeless tobacco within 4 weeks prior to Screening or during the course of the study.
5. Patient has been diagnosed with hairy leukoplakia.
6. Patient has evidence of a systemic infection or has used systemic antibiotics within 14 days prior to start of dosing for males and females of non-childbearing potential or within 30 days prior to start of dosing for Women of Childbearing Potential (WOCBP).
7. Patient is currently taking high doses of vitamin A (> 25,000 USP units per day) or has previously used isotretinoin for the treatment of another condition within 6 months of Screening.
8. Patient is currently taking phenytoin or other prohibited medication
9. Patient's index lesion is a recurrent dysplastic lesion in a previously treated area for oral cancer (previous treatment, bed/excision, etc.).
10. The patient has received radiation or chemoradiation therapy to oral cavity within 2 years of Randomization.
11. The patient has any immune compromising conditions at Screening (i.e. HIV, SLE, etc.) or has been treated with immunomodulating medications within 6 months of Screening.
12. Patient currently has poorly controlled diabetes mellitus (uninterrupted hemoglobin A1c >9% for ≥1 year despite standard care).
13. Patient has a history of cardiac, hepatic (ALT and or AST >2x ULN, Total bilirubin >1.5x ULN at Visit 1), or renal disease (eGFR<45 ml/min/1.73 m2) that, in the opinion of the Investigator, might put the patient at undue risk by participating in the study or interferes with the study drug application or the study assessments.
14. Patient has a history of sensitivity to any of the active ingredients in the study drug (e.g. isotretinoin, propylene glycol, natural mint), or retinoids, or vitamin A.
15. Patient has used oral isotretinoin within 14 days of Screening. Patients must agree to abstain from using oral isotretinoin throughout the duration in the study.
16. Patient has participated in an investigational drug trial in which administration of an investigational study drug occurred within 30 days prior to Randomization.
17. Patient is, in the opinion of the Investigator, not an appropriate candidate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Percentages of patients with overall response will be summarized by treatment | 13 weeks
  Overall response is defined as complete or partial response in either clinical or histological outcome without worsening of either.
The percentages of patients reporting any treatment-emergent adverse event (AE) will be tabulated by system organ class and preferred term for each treatment | 13 weeks

SECONDARY OUTCOMES:
Plasma concentrations of isotretinoin will be summarized by treatment using descriptive statistics | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joy Schleyer, Study Director — Skyline Biosciences
Locations (5):
- United States (5):
  - University of Alabama at Birmingham (UAB) - The Kirklin Clinic (TKC), Birmingham, Alabama
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Carolinas Center for Oral Health, Charlotte, North Carolina
  - PennState Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center - Oral & Maxillofacial Surgery Clinic, Dallas, Texas